CLINICAL TRIAL: NCT05738746
Title: The Effects of the Anti-inflammatory Microbe - Pasteurized Akkermansia Muciniphila (PAM) on Symptoms of Somatic and Mental Stress in Healthcare Professionals
Brief Title: The Efficacy of Pasteurised Akkermansia Muciniphila in Healthy Medical Workers
Acronym: MENTAkHEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: SANPROBI SPOLKA Z OGRANICZONA ODPOWIEDZIALNOSCIA SPOLKA KOMANDYTOWA (Unknown); THE AKKERMANSIA COMPANY (Unknown); Charite University, Berlin, Germany (Other); MAX DELBRUECK CENTRUM FUER MOLEKULARE MEDIZIN IN DER HELMHOLTZ-GEMEINSCHAFT (MDC) - MDC (Unknown); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 101095540
Record Dates: First submitted 2023-01-30; First posted 2023-02-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Stress; Healthy; Dietary Supplement
Keywords: microbiota; postbiotic; stress; metabolome; immunometabolism

STUDY DESIGN:
Intervention Model Description: parallel-groups, randomized, placebo-controlled clinical study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sequentially numbered drug containers of identical appearance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pasteurized Akkermansia muciniphila (Experimental): pasteurized A.muciniphila (Pasteurized, 3x10^10 bacteria per day) as supplement for 3 months,
  Interventions: Dietary Supplement: Pasteurized Akkermansia muciniphila
- Placebo (Placebo Comparator): placebo administered for 3 months once a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pasteurized Akkermansia muciniphila — PAM supplementation; packaging will be given to the subjects every one month during follow-up visits, with the instructions to take one dose every morning on an empty stomach
  Other Names: PAM
  Arms: Pasteurized Akkermansia muciniphila
Dietary Supplement: Placebo — PBO administration; packaging will be given to the subjects every one month during follow-up visits, with the instructions to take one dose every morning on an empty stomach
  Other Names: PBO
  Arms: Placebo

SUMMARY:
Gut microbiota alterations secondary to chronic stress might serve as a triggering factor towards manifestation of somatic and mental symptoms. The administration of pasteurised A. muciniphila MucT has the capability of supporting microbiota and improving the gut barrier integrity, which might lead to decrease of inflammation and the negative health consequences of stress in healthy participants.

DETAILED DESCRIPTION:
The Gut-brain-microbiota axis (GBMA) is a bi-directional pathway, both neuronal and biochemical, between the intestine and the Central Nervous System (CNS). The gut microbiota plays a central role in gut-brain communication. The composition of intestinal microbiota and its functions play an important role in the pathogenesis of disorders of gut-brain interaction - both within the digestive tract and in the brain.

Modulation of gut microbiota with the aid of probiotics, antibiotics, or germ-free feeding protocols significantly altered stressful event-induced behavioral outcomes in rodents. Moreover, the intake of various probiotics significantly improved stress-induced anxiety and depressive-like behaviors in mice. In humans, probiotics were also documented to display some beneficial effects on mental health, including alteration of emotional bias in healthy individuals, and alleviating stress and anxiety among stressed adults.

Psychobiotics are imposed with certain limitations related to their standardization and end-shelf-life product stability. Therefore, the use of postbiotics, which contain bacterial metabolites or other bacteria derived fragments are viewed as novel solutions and alternatives to use of standard probiotics. One of novel postbiotics of interest among scientists and clinicians is pasteurized Akkermansia muciniphila MucT (PAM).

Animal studies indicate that administration of Akkermansia muciniphila can ameliorate metabolic syndrome, obesity, diabetes, and inflammatory bowel disease in animals and has psychobiotic potential. Similar to live A. muciniphila, PAM could ameliorate several diseases as well. The mechanism of action of PAM - improving gut barrier integrity - suggests the potential use to reduce the negative effects of stress. Human studies shown that PAM is safety, what was confirmed in the Scientific Opinion of EFSA. Recently A. muciniphila was approved as the Novel Food.

A proof of concept study will be conducted to verify the hypothesis that PAM reduces the psychological and somatic effects of stress.

ELIGIBILITY:
Inclusion Criteria:

* Working in a high stress hospital department, like: emergency, trauma, intensive care, surgery, internal diseases;
* Written informed consent to participate in this study before any study-mandated procedure;
* Body mass index (BMI) ≥18.5 kg/m2 and ≤ 35 kg/m2;
* A willingness and motivation to follow the study protocol.

Exclusion Criteria:

* Diagnosis of autoimmune, neurological, immunocompromised, thyroid, inflammatory bowel diseases, irritable bowel syndrome, diabetes, cancer, and/or IgE-dependent allergy;
* Psychiatric comorbidities, including mental retardation, organic brain dysfunction, or addiction (except nicotine and caffeine), intake of antipsychotic and antidepressive drugs;
* Proton pump inhibitors usage;
* The use of antibiotics and/or probiotics 4 weeks prior to the study;
* Glucocorticosteroids and/or metformin treatment;
* Dietary supplementation (except for vitamin D) within the three months before screening;
* Specific restrictive (e.g. elimination, vegan, FODMAP, reduction) diet within the three months before screening;
* Significant changes in physical activity 4 weeks before the trial entry;
* Pregnancy or lactation;
* Significant GI surgery within the last 6 months prior to or planned during the study;
* Any other medication for management of IBS complaints like peppermint oil, bile acid binders;
* Lactose intolerance;
* Participation in another study during the last 30 days prior to and during the study;
* Any other reason for exclusion as per investigator's judgment, e.g. insufficient compliance with study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Stress intensity | baseline
  serum dehydroepiandrosterone sulfate (DHEAS) in blood
Stress intensity | 1 month
  serum dehydroepiandrosterone sulfate (DHEAS) in blood
Stress intensity | 3 months
  serum dehydroepiandrosterone sulfate (DHEAS) in blood
Cardiovascular marker of stressor intensity | baseline
  blood pressure
Cardiovascular marker of stressor intensity | 1 month
  blood pressure
Cardiovascular marker of stressor intensity | 3 months
  blood pressure
Cardiovascular marker of stressor intensity | baseline
  heart rate
Cardiovascular marker of stressor intensity | 1 month
  heart rate
Cardiovascular marker of stressor intensity | 3 months
  heart rate
Stress intensity | baseline
  Perceived Stress Scale (PSS-10). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Stress intensity | 1 month
  Perceived Stress Scale (PSS-10). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Stress intensity | 3 months
  Perceived Stress Scale (PSS-10). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Psychosocial working conditions | baseline
  Copenhagen Psychosocial Questionnaire (COPSOQ). The scales of the COPSOQ are formed by adding the points of the individual questions of the scales by giving equal weights to each question. In most cases the questions have five response options. In these cases the weights are: 0, 25, 50, 75, and 100. The scale value is calculated as the simple average
Psychosocial working conditions | 1 month
  Copenhagen Psychosocial Questionnaire (COPSOQ). The scales of the COPSOQ are formed by adding the points of the individual questions of the scales by giving equal weights to each question. In most cases the questions have five response options. In these cases the weights are: 0, 25, 50, 75, and 100. The scale value is calculated as the simple average
Psychosocial working conditions | 3 months
  Copenhagen Psychosocial Questionnaire (COPSOQ). The scales of the COPSOQ are formed by adding the points of the individual questions of the scales by giving equal weights to each question. In most cases the questions have five response options. In these cases the weights are: 0, 25, 50, 75, and 100. The scale value is calculated as the simple average
The recognition of the most common mental disorders | baseline
  Primary Care Evaluation of Mental Disorders (PRIME-MD). The yes/no questionnaire serves as an initial screen for 5 general groups of mental disorders commonly found in the general population
The recognition of the most common mental disorders | 1 month
  Primary Care Evaluation of Mental Disorders (PRIME-MD). The yes/no questionnaire serves as an initial screen for 5 general groups of mental disorders commonly found in the general population
The recognition of the most common mental disorders | 3 months
  Primary Care Evaluation of Mental Disorders (PRIME-MD). The yes/no questionnaire serves as an initial screen for 5 general groups of mental disorders commonly found in the general population
Depression | baseline
  Patient Health Questionnaire-9 (PHQ-9). Nine items, each of which is scored 0 to 3, providing a 0 to 27 severity score.This score can then be referred to the accompanying PHQ-9 Scoring Box to interpret the TOTAL score.
Depression | 1 month
  Patient Health Questionnaire-9 (PHQ-9). Nine items, each of which is scored 0 to 3, providing a 0 to 27 severity score.This score can then be referred to the accompanying PHQ-9 Scoring Box to interpret the TOTAL score.
Depression | 3 months
  Patient Health Questionnaire-9 (PHQ-9). Nine items, each of which is scored 0 to 3, providing a 0 to 27 severity score.This score can then be referred to the accompanying PHQ-9 Scoring Box to interpret the TOTAL score.
Depressive state | baseline
  The Beck Depression Inventory (BDI). When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows:
  0-18: indicates minimal depression 18-30: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
Depressive state | 1 month
  The Beck Depression Inventory (BDI). When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows:
  0-18: indicates minimal depression 18-30: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
Depressive state | 3 months
  The Beck Depression Inventory (BDI). When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows:
  0-18: indicates minimal depression 18-30: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
Anxiety and stress | baseline
  Depression Anxiety Stress Scale 21 (DASS-21). This is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. The rating scale is as follows:
  0 - Did not apply to me at all
  1. - Applied to me to some degree, or some of the time
  2. - Applied to me to a considerable degree, or a good part of time
  3. - Applied to me very much, or most of the time.
  SUBSCALES:
  DASS_Anxiety = questions 2 + 4 + 7 + 9 + 15 + 19 + 20
  DASS_Depression = questions 3 + 5 + 10 + 13 + 16 + 17 + 21
  DASS_Stress = questions 1 + 6 + 8 + 11 + 12 + 14 +18
Anxiety and stress | 1 month
  Depression Anxiety Stress Scale 21 (DASS-21). This is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. The rating scale is as follows:
  0 - Did not apply to me at all
  1. - Applied to me to some degree, or some of the time
  2. - Applied to me to a considerable degree, or a good part of time
  3. - Applied to me very much, or most of the time.
  SUBSCALES:
  DASS_Anxiety = questions 2 + 4 + 7 + 9 + 15 + 19 + 20
  DASS_Depression = questions 3 + 5 + 10 + 13 + 16 + 17 + 21
  DASS_Stress = questions 1 + 6 + 8 + 11 + 12 + 14 +18
Anxiety and stress | 3 months
  Depression Anxiety Stress Scale 21 (DASS-21). This is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. The rating scale is as follows:
  0 - Did not apply to me at all
  1. - Applied to me to some degree, or some of the time
  2. - Applied to me to a considerable degree, or a good part of time
  3. - Applied to me very much, or most of the time.
  SUBSCALES:
  DASS_Anxiety = questions 2 + 4 + 7 + 9 + 15 + 19 + 20
  DASS_Depression = questions 3 + 5 + 10 + 13 + 16 + 17 + 21
  DASS_Stress = questions 1 + 6 + 8 + 11 + 12 + 14 +18
Occurrence of Irritable Bowel Syndrome | baseline
  Rome IV criteria
Occurrence of Irritable Bowel Syndrome | 1 month
  Rome IV criteria
Occurrence of Irritable Bowel Syndrome | 3 months
  Rome IV criteria
Occurence and severity of gastrointestinal symptoms | baseline
  Gastrointestinal Symptom Rating Scale (GSRS)
Occurence and severity of gastrointestinal symptoms | 1 month
  Gastrointestinal Symptom Rating Scale (GSRS)
Occurence and severity of gastrointestinal symptoms | 3 months
  Gastrointestinal Symptom Rating Scale (GSRS)

SECONDARY OUTCOMES:
Microbiota composition | baseline
  next generation sequencing
Microbiota composition | 1 month
  next generation sequencing
Microbiota composition | 3 months
  next generation sequencing
A. muciniphila count in stool | baseline
  real-time quantitative PCR (qPCR)
A. muciniphila count in stool | 1 month
  real-time quantitative PCR (qPCR)
A. muciniphila count in stool | 3 months
  real-time quantitative PCR (qPCR)
Total bacteria count in stool | baseline
  real-time quantitative PCR (qPCR)
Total bacteria count in stool | 1 month
  real-time quantitative PCR (qPCR)
Total bacteria count in stool | 3 months
  real-time quantitative PCR (qPCR)
Short chain fatty acids content in stool | baseline
  quadrupole mass spectrometer and high performance liquid chromatograph
Short chain fatty acids content in stool | 1 month
  quadrupole mass spectrometer and high performance liquid chromatograph
Short chain fatty acids content in stool | 3 months
  quadrupole mass spectrometer and high performance liquid chromatograph
Immune phenotypes of peripheral blood mononuclear cells (PBMCs) | baseline
  single-cell genomics (scRNA-seq and scATAC-seq) analyses (in blood)
Immune phenotypes of peripheral blood mononuclear cells (PBMCs) | 1 month
  single-cell genomics (scRNA-seq and scATAC-seq) analyses (in blood)
Immune phenotypes of peripheral blood mononuclear cells (PBMCs) | 3 months
  single-cell genomics (scRNA-seq and scATAC-seq) analyses (in blood)
Inflammatory mediators concentrations in blood | baseline
  high-throughput protein biomarker analysis with the advent of Proximity Extension Assay
Inflammatory mediators concentrations in blood | 1 month
  high-throughput protein biomarker analysis with the advent of Proximity Extension Assay
Inflammatory mediators concentrations in blood | 3 months
  high-throughput protein biomarker analysis with the advent of Proximity Extension Assay
Zonulin concentration in stool | baseline
  enzyme-linked immunosorbent assay (ELISA)
Zonulin concentration in stool | 1 month
  enzyme-linked immunosorbent assay (ELISA)
Zonulin concentration in stool | 3 months
  enzyme-linked immunosorbent assay (ELISA)
Calprotectin concentration in stool | baseline
  enzyme-linked immunosorbent assay (ELISA)
Calprotectin concentration in stool | 1 month
  enzyme-linked immunosorbent assay (ELISA)
Calprotectin concentration in stool | 3 months
  enzyme-linked immunosorbent assay (ELISA)
Lipopolysaccharide concentration in blood | baseline
  enzyme-linked immunosorbent assay (ELISA)
Lipopolysaccharide concentration in blood | 1 month
  enzyme-linked immunosorbent assay (ELISA)
Lipopolysaccharide concentration in blood | 3 months
  enzyme-linked immunosorbent assay (ELISA)
Adiposity | baseline
  Fat mass/fat free mass evaluated by bioimpedance
Adiposity | 1 month
  Fat mass/fat free mass evaluated by bioimpedance
Adiposity | 3 months
  Fat mass/fat free mass evaluated by bioimpedance
Obesity | baseline
  Body weight
Obesity | 1 month
  Body weight
Obesity | 3 months
  Body weight
Dietary habits | baseline
  the frequency of certain food consumption (rank score) by means of validated Food Frequency Questionnaire (FFQ).
Physical activity | baseline
  International Physical Activity Questionnaire. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week).
Functions of peripheral blood mononuclear cells (PBMCs) | baseline
  mass cytometry (CyTOF)
Functions of peripheral blood mononuclear cells (PBMCs) | 1 month
  mass cytometry (CyTOF)
Functions of peripheral blood mononuclear cells (PBMCs) | 3 months
  mass cytometry (CyTOF)
Insulin resistance | baseline
  HOMA-Homeostasis Model Assessment calculated from fasted glycemia and insulinemia
Insulin resistance | 1 month
  HOMA-Homeostasis Model Assessment calculated from fasted glycemia and insulinemia
Insulin resistance | 3 months
  HOMA-Homeostasis Model Assessment calculated from fasted glycemia and insulinemia
carbohydrate metabolism | baseline
  glycated hemoglobin (HbA1c)
carbohydrate metabolism | 1 month
  glycated hemoglobin (HbA1c)
carbohydrate metabolism | 3 months
  glycated hemoglobin (HbA1c)
Concentration of blood lipids | baseline
  Analysis of circulating lipids : total, LDL and HDL cholesterol (mg/dl), triglycerides (md/dl)
Concentration of blood lipids | 1 month
  Analysis of circulating lipids : total, LDL and HDL cholesterol (mg/dl), triglycerides (md/dl)
Concentration of blood lipids | 3 months
  Analysis of circulating lipids : total, LDL and HDL cholesterol (mg/dl), triglycerides (md/dl)

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Pomeranian Medical University in Szczecin, Szczecin, West Pomeranian Voivodeship
  - Center fo Medical Simulation, Szczecin, West Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided
1. Personal data will be pseudonymised and encrypted, and after the purpose of processing has ceased to exist, they will be deleted or made anonymous.
  2. Personal data will be processed in compliance with the technical and organizational measures referred to in Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 and the Data Protection Policy at PMU.
  3. Research data will be made available in the open research data repository, at the latest when the research article is published, after the end of its analysis.
  4. There are no restrictions or obstacles preventing full disclosure of data.
  5. Sharing data requires no consent of the study participants as for the anonymous character of the study
  6. Only data from sequencing analyzes will be stored indefinitely in the repository https://qiita.ucsd.edu/
  7. The remaining data will be deposited for a minimum of 10 years in the ZENODO repository

REFERENCES:
- [Background] Depommier C, Everard A, Druart C, Plovier H, Van Hul M, Vieira-Silva S, Falony G, Raes J, Maiter D, Delzenne NM, de Barsy M, Loumaye A, Hermans MP, Thissen JP, de Vos WM, Cani PD. Supplementation with Akkermansia muciniphila in overweight and obese human volunteers: a proof-of-concept exploratory study. Nat Med. 2019 Jul;25(7):1096-1103. doi: 10.1038/s41591-019-0495-2. Epub 2019 Jul 1. PMID 31263284
- [Background] Schneeberger M, Everard A, Gomez-Valades AG, Matamoros S, Ramirez S, Delzenne NM, Gomis R, Claret M, Cani PD. Akkermansia muciniphila inversely correlates with the onset of inflammation, altered adipose tissue metabolism and metabolic disorders during obesity in mice. Sci Rep. 2015 Nov 13;5:16643. doi: 10.1038/srep16643. PMID 26563823
- [Background] Druart C, Plovier H, Van Hul M, Brient A, Phipps KR, de Vos WM, Cani PD. Toxicological safety evaluation of pasteurized Akkermansia muciniphila. J Appl Toxicol. 2021 Feb;41(2):276-290. doi: 10.1002/jat.4044. Epub 2020 Jul 28. PMID 32725676
- [Background] Cani PD, Depommier C, Derrien M, Everard A, de Vos WM. Akkermansia muciniphila: paradigm for next-generation beneficial microorganisms. Nat Rev Gastroenterol Hepatol. 2022 Oct;19(10):625-637. doi: 10.1038/s41575-022-00631-9. Epub 2022 May 31. PMID 35641786
- See also: EC official website with research results — http://cordis.europa.eu/project/id/101095540